CLINICAL TRIAL: NCT03585179
Title: Oral and 5% Topical Tranexamic Acid in Monotherapy Compared With 4% Topical Hydroquinone for the Treatment of Melasma: Three-arm Randomized, Double-blinded Clinical Trial
Brief Title: Oral and Topical Tranexamic Acid for the Treatment of Melasma
Acronym: TRANEXAMICO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centro Dermatológico Dr. Ladislao de la Pascua (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 151/2018
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Melasma; Chloasma; Melanosis
Keywords: Melasma; Chloasma; Melanosis; Tranexamic acid; Hydroquinone; Therapeutics
MeSH Terms: conditions — Melanosis | interventions — Tranexamic Acid; hydroquinone

STUDY DESIGN:
Intervention Model Description: Three-arm clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will receive both topical and oral interventions. Group 1: pills of tranexamic acid 250 mg bid plus placebo gel bid, Group 2: pills of placebo bid plus 5% tranexamic acid gel bid and Group 3: pills of placebo bid plus 4% hydroquinone cream at night and a placebo cream at morning. Containers will be of identical appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Oral tranexamic acid (Experimental): 250 mg of tranexamic acid bid orally
  Interventions: Drug: Oral Tranexamic Acid
- Topical tranexamic acid (Experimental): 5% topical tranexamic acid bid
  Interventions: Drug: 5% topical tranexamic acid
- Topical hydroquinone (Active Comparator): 4% hydroquinone once daily at night
  Interventions: Drug: 4% hydroquinone

INTERVENTIONS:
Drug: Oral Tranexamic Acid — Participants will take a pill of 250 mg bid for 12 weeks
  Arms: Oral tranexamic acid
Drug: 5% topical tranexamic acid — Participants will apply a layer of gel on the affected skin bid for 12 weeks
  Other Names: Topical tranexamic acid
  Arms: Topical tranexamic acid
Drug: 4% hydroquinone — Participants will apply a layer of cream on the affected skin once at night
  Other Names: Hydroquinone
  Arms: Topical hydroquinone

SUMMARY:
Tranexamic acid has been used for treating melasma due to its effect on decreasing the activity of tyrosinase and melanogenesis. This 3-arm clinical trial will asess the efficacy and safety of oral and topical tranexamic acid as monotherapy compared with topical hydroquinone for 12 weeks in adults with melasma. The primary outcome will be the percentage of reduction at 12-week period of mMASI and melanin index. The incidence of adverse effects will be reported at weeks 4, 8 and 12.

DETAILED DESCRIPTION:
Tranexamic acid has been used for treating melasma due to its effect on decreasing the activity of tyrosinase and melanogenesis. This 3-arm clinical trial will asess the efficacy and safety of oral and topical tranexamic acid as monotherapy compared with topical hydroquinone for 12 weeks in adults with melasma. One hundred and twenty patients will be recruited in 3 groups of intervention: group I with tranexamic acid at a dose of 250 mg bid orally, group II with 5% topical tranexamic acid bid, group III with 4% topical hydroquinone once daily. The primary outcome will be the percentage of reduction at 12-week period of mMASI and melanin index. The incidence of adverse effects will be reported at weeks 4, 8 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* Moderate to severe melasma
* History of multiple topical depigmenting treatments and use of photoprotection, with subjective improvement less than 50% or mMASI <50% reported by the dermatologist after one year of treatment.

Exclusion Criteria:

* Pregnancy
* Hormonal contraception
* Lactation
* Treatment with hydroquinone or tranexamic acid at the time of the study or in the last 3 months
* Endocrinology diseases
* Hormone replacement therapy
* Family or personal history of one of the following: autoimmune disorders, coagulation disorders, chronic venous insufficiency, heart diseases, retinopathies, kidney disorders
* Mental disability

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Change of mMASI (Modified Melasma Area and Severity Index) | 12 weeks
  The difference between mMASI (Modified Melasma Area and Severity Index) at week 0 and mMASI (Modified Melasma Area and Severity Index) at week 12

SECONDARY OUTCOMES:
Change in Quality of life | 12 weeks
  The reported change of the score of DLQI (Dermatology Life Quality Index) at week 0 versus week 12. Total score ranges from 0 to 30 and the difference between the score at week 0 and week 12 will be calculated.
Melanin index | 12 weeks
  The difference between melanin index at week 0 versus week 12. The melanin index will be measure with Mexameter® MX 18. Total index ranges from 0 to 999.

CONTACTS AND LOCATIONS:
Overall Officials: Martha A Morales-Sánchez, MD, Study Director — Centro Dermatológico Dr. Ladislao de la Pascua
Locations (1):
- Centro Dermatológico "Dr. Ladislao de la Pascua", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
Only if researchers ask for the complete data of the trial.